CLINICAL TRIAL: NCT01965860
Title: The Study of Transferability and Cost-effectiveness of a Proficiency-based Stepwise Endovascular Curricular Training Program (PROSPECT) in Surgical Trainees
Brief Title: Transferability and Cost-effectiveness of PROSPECT in Surgical Trainees
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013/783
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-01

CONDITIONS: Vascular Disease
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Initially 39 participants were enrolled, 7 excluded because they declined to participate. 32 people were randomized.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PROSPECT (Experimental): the trainee will study four modules of E-learning (basic endovascular skills module, iliac artery module, superficial femoral artery module and postoperative care module). After studying each module the trainee will complete a Multiple Choice Questionnaire and perform a simple and a complex exercise on the simulator.
  Interventions: Other: additional curriculum (E-learning + simulation)
- CONTROL (No Intervention): The trainee will continue clinical education without additional curriculum, but will be allowed to study independently.
- E-LEARNING (Experimental): the trainee will study four modules of E-learning (basic endovascular skills module, iliac artery module, superficial femoral artery module and postoperative care module). After studying each module the trainee will complete a Multiple Choice Questionnaire, no simulation.
  Interventions: Other: additional E-learning

INTERVENTIONS:
Other: additional curriculum (E-learning + simulation)
  Arms: PROSPECT
Other: additional E-learning
  Arms: E-LEARNING

SUMMARY:
To design, validate and prove cost-effectiveness of a comprehensive endovascular simulation curriculum consisting of cognitive and psychomotor skills training for endovascular management of symptomatic vascular disease in the lower limbs.

DETAILED DESCRIPTION:
The main goal is to design a comprehensive endovascular simulation curriculum consisting of cognitive and psychomotor skills training for endovascular management of symptomatic vascular disease in the lower limbs (Rutherford classification 2-5; stenosis or occlusion in the iliac, superficial femoral and popliteal arteries). The curriculum will consist of E-learning, video-based learning and simulation exercises on the Virtual Reality simulator on which an endovascular procedure will be simulated.

Skills transferability to real life practice will be verified by means of a RCT. In this RCT the investigators will compare the cognitive knowledge and technical performance of curricular trained surgical trainees with conventionally trained trainees during treatment of patients under supervision. The hypothesis states that surgeons trained within the PROSPECT curriculum will show improved technical knowledge of endovascular treatment of atherosclerotic disease in the iliac, superficial femoral and popliteal arteries and will demonstrate increased technical proficiency in the angiosuite in comparison with surgeons who received only conventional training. Subjects will be surgical trainees (N=32). They will be randomized into a three groups: a control group (N=11), a group that only has access to E-learning (N=10) and a PROSPECT group (N=11). Both groups will continue their traditional clinical education and the PROSPECT group will additionally be trained within this endovascular curriculum. The investigators hope that this study may ultimately lead to an improvement in the quality of patient care by standardizing competencies of endovascular operators in training and practice.

Additionally a cost-effectiveness analysis of PROSPECT compared to traditional training modalities will be executed. A successful training program is expected to lead to a shortening of the learning curve, reduction in number of errors during real life procedures and more efficient use of hybrid angio suites. The financial impact of potentially shorter duration of endovascular interventions will be studied and compared to time investment and additional costs associated with stepwise, supervised training using VR simulators.

ELIGIBILITY:
Inclusion Criteria:

* Surgical trainee
* Knowledge and technical skill level evaluated
* Demographics questionnaire and general MCQ test completed
* 2 endovascular simulated exercises completed after familiarization with the simulator

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Van Herzeele, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Background] Maertens H, Aggarwal R, Desender L, Vermassen F, Van Herzeele I. Development of a PROficiency-Based StePwise Endovascular Curricular Training (PROSPECT) Program. J Surg Educ. 2016 Jan-Feb;73(1):51-60. doi: 10.1016/j.jsurg.2015.07.009. Epub 2015 Aug 11. PMID 26276301
- [Result] Maertens H, Aggarwal R, Moreels N, Vermassen F, Van Herzeele I. A Proficiency Based Stepwise Endovascular Curricular Training (PROSPECT) Program Enhances Operative Performance in Real Life: A Randomised Controlled Trial. Eur J Vasc Endovasc Surg. 2017 Sep;54(3):387-396. doi: 10.1016/j.ejvs.2017.06.011. Epub 2017 Jul 19. PMID 28734705
- [Result] Maertens H, Vermassen F, Aggarwal R, Doyen B, Desender L, Van Herzeele I, Annemans L. Endovascular Training Using a Simulation Based Curriculum is Less Expensive than Training in the Hybrid Angiosuite. Eur J Vasc Endovasc Surg. 2018 Oct;56(4):583-590. doi: 10.1016/j.ejvs.2018.07.011. Epub 2018 Aug 18. PMID 30131277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for RCT (before 02/2016): general surgery trainees from Ghent University Recruitment for registry (after 02/2016): general surgery trainees from Ghent University, Leuven University, Nancy University, Lille University, CAMES Copenhagen
Pre-assignment Details: 7 people declined to participate before randomisation during the RCT
Groups:
- PROSPECT: the trainee will study four modules of E-learning (basic endovascular skills module, iliac artery module, superficial femoral artery module and postoperative care module. After studying each module the trainee will complete a Multiple Choice Questionnaire and perform a simple and a complex exercise on the simulator.
  additional curriculum
- E-LEARNING: the trainee will study four modules of E-learning (basic endovascular skills module, iliac artery module, superficial femoral artery module and postoperative care module. After studying each module the trainee will complete a Multiple Choice Questionnaire. No simulation exercises.
Period: Overall Study
Arm/Group | PROSPECT | E-LEARNING | CONTROL
Started | 11 | 10 | 11
Completed | 9 | 10 | 10
Not Completed | 2 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Logistics | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 39 surgical trainees were eligible to start the RCT. Randomisation took place after screening for eligibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | PROSPECT | E-LEARNING | CONTROL | Total
Number analyzed (Participants) | 11 | 10 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants] — Population: Row population differs from overall as participants are spread accross study arms.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 11 | 10 | 11 | 32
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants are spread accross study arms.
  Participants
    Female | 5 | 6 | 5 | 16
    Male | 6 | 4 | 6 | 16
Postgraduate year [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants are spread accross study arms
  Participants
    Level 1 | 2 | 3 | 4 | 9
    Level 2 | 2 | 3 | 1 | 6
    Level 3 | 4 | 1 | 3 | 8
    Level 4 | 0 | 2 | 1 | 3
    Level 5 | 1 | 1 | 1 | 3
    Level 6 | 2 | 0 | 1 | 3
No. endovascular cases assisted [Count of Participants; unit: Participants] — Population: Row population differs from the overall as participants are spread accross study arms
  Participants
    0-5 | 1 | 2 | 2 | 5
    5-10 | 2 | 1 | 1 | 4
    10-50 | 6 | 5 | 1 | 12
    50-100 | 1 | 1 | 5 | 7
    100-200 | 1 | 0 | 0 | 1
    > 200 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Technical and Global Performance of the Surgical Trainee in Real Life Procedures
Description: The consultant will assess the trainee during the intervention.
  * Global Rating Scale of Endovascular Performance (Range 11-55): to rate the global performance - modified OSATS (Objective Structured Assessment of Technical Skills) scale
  * Examiner Checklist for Diagnostic Angiography, Angioplasty and Stenting (Range 17-85): to rate the technical performance
  For both scales, the higher the score, the better. Surrogate measures of performance are also evaluated (total procedure and fluoroscopy time, radiation dose, contrast volume and number of endovascular tools used). Post-hoc videos of hand movements and the fluoroscopy imaging recorded during the real procedure will be rated using the same scoring systems. Two real life endovascular procedures will be performed within six weeks after completing the curriculum. Evaluation will occur during the intervention and videos of hand movements and fluoroscopy imaging will be evaluated afterwards.
Time Frame: 6 weeks after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROSPECT | E-LEARNING | CONTROL
Number analyzed (Participants) | 9 | 10 | 10
score on a scale
  GRS (real life simulation) | 39.36 (2.05) | 28.42 (2.15) | 23.09 (2.18)
  Checklist (real life simulation) | 63.51 (3.18) | 53.63 (3.34) | 38.72 (3.38)

2. Secondary Outcome: Improved Knowledge and Technical Performance of the Surgical Trainee on a Simulated Complex Module
Description: The cognitive and technical skills retention of the surgical trainee is measured by a MCQ test and a simulation based exercise, pre and post PROSPECT.
  MCQ test: validated Multiple Choice Test - Range 0-20 GRS: Global Rating Scale of Endovascular Performance, modified OSATS (Objective Structured Assessment of Technical Skills) scale: to assess global performance (same as primary outcome) - Range: 11-55 Examiners checklist: Examiner Checklist for Diagnostic Angiography, Angioplasty and Stenting: to assess technical performance (same as primary objective) - Range: 17-85
  For al outcome measures: the higher the score, the better
Time Frame: Pre curriculum, 6 weeks and 3 months after completion of the curriculum (3 months only for intervention arms)
Measure: Mean (Standard Deviation); unit: score on a test or scale
Arm/Group | PROSPECT | E-LEARNING | CONTROL
Number analyzed (Participants) | 9 | 10 | 10
score on a test or scale
  Pre-test MCQ | 14 (3.39) | 14.88 (1.13) | 14 (2.49)
  Post test MCQ 6w | 18.11 (1.36) | 17.88 (0.99) | 15.2 (2.7)
  Post test MCQ 3m | 18.25 (1.98) | 17.71 (0.75) | NA (NA) — data not collected from this arm/group at 3m
  Pre GRS | 19.78 (7.24) | 16.25 (4.1) | 18 (7.75)
  Post GRS 6w | 49.56 (3.78) | 32.75 (13.51) | 21.2 (7.48)
  Post GRS 3m | 51.13 (3.44) | 24.14 (6.65) | NA (NA) — data not collected from this arm/group at 3m
  Pre Examiner Checklist | 43.56 (15.76) | 35.63 (11.38) | 37.6 (13.98)
  Post Examiner Checklist 6w | 83.22 (1.99) | 59.25 (16.73) | 42.8 (15.39)
  Post Examiner Checklist 3m | 82.25 (1.75) | 51.71 (16.31) | NA (NA) — data not collected from this arm/group at 3m
Statistical Analysis 1: Comparison: PROSPECT vs E-LEARNING vs CONTROL; Prior to the study a power analysis was performed to calculate the number of participants required in each of the three groups. Previous work comparing OSATS derived scores in endovascular interventions shows a Cohen D of two. Using a of .05, a power of .80, and an expected dropout rate of 10%, the minimum number of surgical trainees required per group was seven. Null hypothesis for primary outcome: no difference in technical performance during real life procedures between the three groups; Test type: Superiority; p = 0.001, ANOVA
Statistical Analysis 2: Comparison: PROSPECT; Null Hypothesis: There is no difference in Pre and Post test MCQ score; Test type: Other; p = 0.003, ANOVA
Statistical Analysis 3: Comparison: E-LEARNING; Null Hypothesis: There is no difference in Pre and Post test MCQ score; Test type: Other; p = 0.001, ANOVA
Statistical Analysis 4: Comparison: CONTROL; Null Hypothesis: There is no difference in Pre and Post test MCQ score; Test type: Other; p = 0.228, ANOVA
Statistical Analysis 5: Comparison: PROSPECT; Null Hypothesis: There is no difference in Pre and Post test GRS score; Test type: Other; p = 0.001, ANOVA
Statistical Analysis 6: Comparison: E-LEARNING; Null Hypothesis: There is no difference in Pre and Post test GRS score; Test type: Other; p = 0.008, ANOVA
Statistical Analysis 7: Comparison: CONTROL; Null Hypothesis: There is no difference in Pre and Post test GRS score; Test type: Other; p = 0.164, ANOVA
Statistical Analysis 8: Comparison: PROSPECT; Null Hypothesis: There is no difference in Pre and Post test Examiner's checklist score; Test type: Other; p = 0.001, ANOVA
Statistical Analysis 9: Comparison: E-LEARNING; Null Hypothesis: There is no difference in Pre and Post test Examiner's checklist score; Test type: Other; p = 0.001, ANOVA
Statistical Analysis 10: Comparison: CONTROL; Null Hypothesis: There is no difference in Pre and Post test Examiner's checklist score; Test type: Other; p = 0.190, ANOVA

3. Other Pre Specified Outcome: PROSPECT Proficiency
Description: After the RCT, a registry was started with all participants that started PROSPECT. Outcome: do PROSPECT participants pass the curriculum, do they become proficient?
Time Frame: After RCT
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Description: Participants were not at risk of adverse events as they were not patients but healthy trainees. There was monitoring/assesment for all-cause mortality, serious and other (not including serious) adverse events, but none occured.
Arm/Group | PROSPECT | E-LEARNING | CONTROL
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
* Single centre, results may not be applicable to other centres/countries.
* Randomisation status was not blinded for participants, consultant can unintentionally know randomisation group.
* Long-term skills retention was not assessed beyond 3 months post-training.
* As the procedures were closely supervised, operative metrics cannot be used to assess the operative performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes